CLINICAL TRIAL: NCT03656978
Title: Ultrasound-Guided Vascular Puncture and Catheterization
Acronym: UGVPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Chunhua Yu, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: zs-1338
Record Dates: First submitted 2018-08-21; First posted 2018-09-04 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Vascular Access Complication; Ultrasound Therapy; Complications; Perioperative/Postoperative Complications; Cardiovascular Abnormalities
Keywords: vascular access; vascular catheterization; ultrasound-guided; ultrasonography; perioperative; anesthesia; cardiovascular abnormalities
MeSH Terms: conditions — Postoperative Complications; Cardiovascular Abnormalities

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dynamic (Active Comparator): Keep moving the probe for needle tip visualization during the puncture procedure.
  Interventions: Behavioral: dynamic
- Regular-triangle (Placebo Comparator): Needle access along the hypotenuse of the regular triangle formed by the vascular depth and puncture point.
  Interventions: Behavioral: Regular-triangle

INTERVENTIONS:
Behavioral: dynamic — Use the according methods in dynamic arm descriptions.
  Arms: Dynamic
Behavioral: Regular-triangle — Use the according methods in regular-triangle arm descriptions.
  Arms: Regular-triangle

SUMMARY:
To assess and improve the safety and success rate of vascular puncture and catheterization using ultrasound-guided methods.

DETAILED DESCRIPTION:
Investigators hypothesized that （1） various ultrasound-guided methods had different performances of vascular puncture and catheterization, (2) certain risk factors influenced safety and success rate of vascular puncture and catheterization (3) implementation of protocols could improve the performances of ultrasound-guided vascular puncture and catheterization.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years old.
* Scheduled for selective surgery.
* Requirement of perioperative vascular puncture and catheterization.
* American standard of anesthesia level I-IV.

Exclusion Criteria:

* Contraindication to vascular puncture or catheterization.
* Occlusion or thrombosis of target vessel evaluated by ultrasound.
* Refuse or disagreement from participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-04-23 (Actual); Study Completion 2019-03-08 (Actual)

PRIMARY OUTCOMES:
Successful rate without extra vascular damage | Through study completion, an average of 1 year.
  Percentages of successful catheterization without vascular damage of posterior wall.

SECONDARY OUTCOMES:
Successful rate at first attempt. | Through study completion, an average of 1 year.
  Percentage of successful catheterization at first attempt without needle withdraw.
Time duration of catheterization. | Through study completion, an average of 1 year.
  From beginning of needle puncture to finishing or failing catheterization.
Relative factors of successful catheterization without posterior wall damage. | Through study completion, an average of 1 year.
  Relationship between independent variables (gender, age, BMI, BP, depth and so on) and successful catheterization without posterior wall damage.
The effect of depth to the successful catheterization without posterior wall puncture. | Through study completion, an average of 1 year.
  The relationships between different depth of vascular anterior wall and successful catheterization without posterior wall puncture.

CONTACTS AND LOCATIONS:
Overall Officials: Yu, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Performances of vascular manufacture，such as posterior wall puncture，success at first attempt， overall success or failure and so on. Evaluations of vascular sonography， such as depth，diameter and so on.

REFERENCES:
- [Background] Sethi S, Maitra S, Saini V, Samra T, Malhotra SK. Comparison of short-axis out-of-plane versus long-axis in-plane ultrasound-guided radial arterial cannulation in adult patients: a randomized controlled trial. J Anesth. 2017 Feb;31(1):89-94. doi: 10.1007/s00540-016-2270-6. Epub 2016 Oct 19. PMID 27761661
- [Background] Goh G, Tan C, Weinberg L. Dynamic ultrasound-guided, short axis, out-of-plane radial artery cannulation: the 'follow the tip' technique. Anaesth Intensive Care. 2013 May;41(3):431-2. No abstract available. PMID 23659411
- [Background] Powell JT, Mink JT, Nomura JT, Levine BJ, Jasani N, Nichols WL, Reed J, Sierzenski PR. Ultrasound-guidance can reduce adverse events during femoral central venous cannulation. J Emerg Med. 2014 Apr;46(4):519-24. doi: 10.1016/j.jemermed.2013.08.023. Epub 2014 Jan 22. PMID 24462032
- [Background] Nakayama Y, Nakajima Y, Sessler DI, Ishii S, Shibasaki M, Ogawa S, Takeshita J, Shime N, Mizobe T. A novel method for ultrasound-guided radial arterial catheterization in pediatric patients. Anesth Analg. 2014 May;118(5):1019-26. doi: 10.1213/ANE.0000000000000164. PMID 24781571
- [Background] Ward F, Faratro R, McQuillan RF. Ultrasound-Guided Cannulation of the Hemodialysis Arteriovenous Access. Semin Dial. 2017 Jul;30(4):319-325. doi: 10.1111/sdi.12603. Epub 2017 May 9. PMID 28486776
- [Background] Fragou M, Gravvanis A, Dimitriou V, Papalois A, Kouraklis G, Karabinis A, Saranteas T, Poularas J, Papanikolaou J, Davlouros P, Labropoulos N, Karakitsos D. Real-time ultrasound-guided subclavian vein cannulation versus the landmark method in critical care patients: a prospective randomized study. Crit Care Med. 2011 Jul;39(7):1607-12. doi: 10.1097/CCM.0b013e318218a1ae. PMID 21494105
- [Background] Reusz G, Csomos A. The role of ultrasound guidance for vascular access. Curr Opin Anaesthesiol. 2015 Dec;28(6):710-6. doi: 10.1097/ACO.0000000000000245. PMID 26539789
- [Background] Gao YB, Yan JH, Ma JM, Liu XN, Dong JY, Sun F, Tang LW, Li J. Effects of long axis in-plane vs short axis out-of-plane techniques during ultrasound-guided vascular access. Am J Emerg Med. 2016 May;34(5):778-83. doi: 10.1016/j.ajem.2015.12.092. Epub 2016 Jan 6. PMID 26830218
- [Derived] Flumignan RL, Trevisani VF, Lopes RD, Baptista-Silva JC, Flumignan CD, Nakano LC. Ultrasound guidance for arterial (other than femoral) catheterisation in adults. Cochrane Database Syst Rev. 2021 Oct 12;10(10):CD013585. doi: 10.1002/14651858.CD013585.pub2. PMID 34637140
- [Derived] Bai B, Tian Y, Zhang Y, Yu C, Huang Y. Dynamic needle tip positioning versus the angle-distance technique for ultrasound-guided radial artery cannulation in adults: a randomized controlled trial. BMC Anesthesiol. 2020 Sep 14;20(1):231. doi: 10.1186/s12871-020-01152-1. PMID 32928119